CLINICAL TRIAL: NCT03058185
Title: Observatoire Des Patients Atteints de Laminopathies et Emerinopathies (Observatory for PAtients With Laminopathies and Emerinopathies)
Acronym: OPALE
Status: Recruiting | Type: Observational
Sponsor: Pitié-Salpêtrière Hospital (Other)
Collaborators: Institute of Myology (Other); Assistance Publique - Hôpitaux de Paris (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Bruno Eymard, Clinical Professor-Neuromuscular Unit, Pitié-Salpêtrière Hospital
Other Study IDs: CPP58-12, ID-RCB2012-A00791
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Laminopathies; Emerinopathies
Keywords: Lamin A/C; LMNA; Emerin; EMD
MeSH Terms: conditions — Laminopathies; X-Linked Emery-Dreifuss Muscular Dystrophy; Autosomal Emery-Dreifuss Muscular Dystrophy; Muscular Dystrophy, Emery-Dreifuss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Laminopathies and emerinopathies are complex group of rare disorders due to mutations in A-type lamins (LMNA) and Emerin (EMD) genes. Among them, disorders affecting skeletal and/or cardiac muscles are the most frequent clinical manifestations, with cardiac disease being a major cause of death. Remarkable progress has been made in the description of the clinical and genetic spectrum of these diseases since the 1990's. Until now, precise phenotype/genotype relations remain elusive. As for several other neuromuscular disorders, apart from symptomatic treatments, there is currently no specific treatment to prevent or slow down the progression of the disease. The OPALE registry is a multicentre web-based registry dedicated to laminopathy and emerinopathy French patients. OPALE has been approved by ethical and regulatory authorities. Its main inclusion criteria is the presence of a proven pathogenic LMNA and/or EMD gene mutation.

The OPALE objectives are to provide a tool allowing detailed capture of patient genetic, neurological, cardiological, endocrinological and respiratory assessments, in order to allow i) precise disease natural history, ii) evaluation of different disease complication frequency and iii) identification of prognosis factors.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a proven pathogenic LMNA and/or EMD gene mutation
* Regular followup in France.
* Signed informed consent

Exclusion Criteria:

-Refusal to sign an informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a proven pathogenic LMNA and/or EMD gene mutation
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-07-11 (Actual); Primary Completion 2033-07-11 (Estimated); Study Completion 2033-07-11 (Estimated)

PRIMARY OUTCOMES:
Comprehensive clinical evaluation of individuals with geneticaly proven mutations in LMNA or EMD genes according to the study protocol, in order to evaluate disease progression | yearly up to 10 years
  Comprehensive clinical evaluation of individuals with geneticaly proven mutations in LMNA or EMD genes according to the study protocol, in order to evaluate disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Karim Wahbi, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Gisele Bonne, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Rabah Ben Yaou, MD, Principal Investigator — Institut de myologie
Locations (28):
- France (28):
  - Centre de référence maladies neuromusculaires,CHU d'Angers, Angers, Angers
  - CHU Strasbourg, Strasbourg, Bas-Rhin
  - CHU Marseille, Marseille, Bouches-du-Rhône
  - CHU Caen, Caen, Calvados
  - CHU Brest, Brest, Finistère
  - CHU Nimes, Nîmes, Gard
  - CHU Bordeaux, Bordeaux, Gironde
  - Centre de Référence de Pathologie NeuroMusculaire, CHU Toulouse, Toulouse, Haute-Garonne
  - CHU Montpelleir, Montpellier, Hérault
  - CHU Rennes, Rennes, Ille-et-Vilaine
  - CHU Tours, Tours, Indre-et-Loire
  - Centre de référence des maladies neuromusculaires, CHRU Lille, Lille, Lille
  - Laboratoire d'Explorations Fonctionnelle, CHU Nantes, Nantes, Loire-Atlantique
  - Centre de référence des maladies neuromusculaires, CHU Lyon, Lyon, Lyon
  - CHU Nancy, Nancy, Meurthe-et-Moselle
  - Centre de référence maladies neuromusculaires ile de France, Hôpital Armand Trousseau, Paris, Paris
  - I-Motion Pédiatrique, Hôpital Armand Trousseau, Paris, Paris
  - Service d'endocrinologie, diabétologie et endocrinologie de la reproduction, Hôpital Saint Antoine, Paris, Paris
  - Centre de référence maladies neuromusculaires ile de France, Institut de myologie, GH Pitié-Salpêtrière, Paris, Paris
  - Institut de cardiologie, GH Pitié-Salpêtrière, Paris, Paris
  - Service de cardiologie, Hôpital Cochin, Paris, Paris
  - Cardiologie et maladies vasculaires, Hôpital Européen Georges-Pompidou HEGP, Paris, Paris
  - CHU Clermont-Ferrand, Clermont-Ferrand, Puy-de-Dôme
  - CHU Rouen, Rouen, Seine-Maritime
  - Centre Expert de Pathologie Neuromusculaire - Département de Pathologie, Créteil, Val-de-Marne
  - Centre de référence des maladies neuromusculaires Ile de France, Hôpital Raymond Poincaré, Garches, Yvelines
  - CHU Grenoble, Grenoble
  - Centre de référence maladies neuromusculaires ile de France, Hôpital Necker Enfants malades, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wahbi K, Ben Yaou R, Gandjbakhch E, Anselme F, Gossios T, Lakdawala NK, Stalens C, Sacher F, Babuty D, Trochu JN, Moubarak G, Savvatis K, Porcher R, Laforet P, Fayssoil A, Marijon E, Stojkovic T, Behin A, Leonard-Louis S, Sole G, Labombarda F, Richard P, Metay C, Quijano-Roy S, Dabaj I, Klug D, Vantyghem MC, Chevalier P, Ambrosi P, Salort E, Sadoul N, Waintraub X, Chikhaoui K, Mabo P, Combes N, Maury P, Sellal JM, Tedrow UB, Kalman JM, Vohra J, Androulakis AFA, Zeppenfeld K, Thompson T, Barnerias C, Becane HM, Bieth E, Boccara F, Bonnet D, Bouhour F, Boule S, Brehin AC, Chapon F, Cintas P, Cuisset JM, Davy JM, De Sandre-Giovannoli A, Demurger F, Desguerre I, Dieterich K, Durigneux J, Echaniz-Laguna A, Eschalier R, Ferreiro A, Ferrer X, Francannet C, Fradin M, Gaborit B, Gay A, Hagege A, Isapof A, Jeru I, Juntas Morales R, Lagrue E, Lamblin N, Lascols O, Laugel V, Lazarus A, Leturcq F, Levy N, Magot A, Manel V, Martins R, Mayer M, Mercier S, Meune C, Michaud M, Minot-Myhie MC, Muchir A, Nadaj-Pakleza A, Pereon Y, Petiot P, Petit F, Praline J, Rollin A, Sabouraud P, Sarret C, Schaeffer S, Taithe F, Tard C, Tiffreau V, Toutain A, Vatier C, Walther-Louvier U, Eymard B, Charron P, Vigouroux C, Bonne G, Kumar S, Elliott P, Duboc D. Development and Validation of a New Risk Prediction Score for Life-Threatening Ventricular Tachyarrhythmias in Laminopathies. Circulation. 2019 Jul 23;140(4):293-302. doi: 10.1161/CIRCULATIONAHA.118.039410. Epub 2019 Jun 3. PMID 31155932
- See also: Portail épidémiologie France — https://epidemiologie-france.aviesan.fr/epidemiologie-france/fiches/observatoire-des-patients-atteints-de-laminopathies-et-emerinopathies
- See also: Orphanet — https://www.orpha.net/en/research-trials/registry/460501?name=Autosomal%20dominant%20Emery-Dreifuss%20muscular%20dystrophy&mode=pat&country=
- See also: AFM-Telethon — https://www.afm-telethon.fr/fr/essais/laminopathie-ou-demerinopathie-lobservatoire-opale